CLINICAL TRIAL: NCT03280667
Title: Denosumab and Pembrolizumab in Clear Cell Renal Carcinoma: a Phase II Trial (ANZUP 1601)
Brief Title: Denosumab and Pembrolizumab in Clear Cell Renal Carcinoma
Acronym: KEYPAD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Australian and New Zealand Urogenital and Prostate Cancer Trials Group (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANZUP1601; 20149171 (Other: Amgen); 53963 (Other: MSD)
Record Dates: First submitted 2017-09-07; First posted 2017-09-12 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-02

CONDITIONS: Renal Cell Carcinoma, Clear Cell; Metastatic Kidney Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — pembrolizumab; Denosumab

STUDY DESIGN:
Intervention Model Description: Single-arm, multicentre, phase 2 trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab plus Denosumab (Experimental): Pembrolizumab 200 mg IV every 3 weeks plus denosumab 120 mg SC on day 1, 8, 22 and then every 3 weeks with daily oral calcium and vitamin D, continued until disease progression or prohibitive toxicity
  Interventions: Drug: Pembrolizumab plus denosumab

INTERVENTIONS:
Drug: Pembrolizumab plus denosumab — Pembrolizumab 200 mg IV every 3 weeks plus denosumab 120 mg SC on day 1, 8, 22 and then every 3 weeks with daily oral calcium and vitamin D
  Other Names: Keytruda and Xgeva

SUMMARY:
This Single-arm, multicentre, phase 2 trial aims determine the activity and safety of pembrolizumab and denosumab in advanced clear cell renal cell carcinoma (ccRCC).

DETAILED DESCRIPTION:
Renal cell carcinoma (RCC) is the 9th most common cancer in Australia, the 10th most common cancer in Western populations1. Approximately 75% of kidney cancers are clear-cell renal cell carcinomas (ccRCC). Current treatments for metastatic ccRCC include VEGFR tyrosine kinase inhibitors (TKIs) and mTOR inhibitors and while many patients benefit from first-line VEGFR TKIs, progression is inevitable and these treatments remain palliative. Second-line VEGFR TKIs and mTOR inhibitors have some benefit but in a smaller increment than first-line treatment. ccRCC is highly immunogenic with benefit from adjuvant autologous vaccines, high-dose IL2 in selected patients and spontaneous remissions seen in a fraction of patients. Cytokine immunotherapy delivered durable complete responses in a subset of patients who survived the very high toxicity of these agents, but use of cytokine immunotherapy is uncommon in modern practice.

Preclinical data and case reports suggest that denosumab, an inhibitor of RANKL signalling, might potentiate the anti-tumour effects of immunotherapy with pembrolizumab, an antibody directed against PD-1, without overlapping toxicities.

This study aims to determine the activity and safety of pembrolizumab and denosumab in advanced clear cell renal cell carcinoma (ccRCC), in patients with disease progression during or after VEGFR TKI treatment.

Adults with unresectable or metastatic ccRCC progressing after treatment with a VEGFR TKI. Key eligibility criteria include target lesion(s) according to RECIST 1.1, good performance status (ECOG PS 0-2), no history of significant autoimmune disease, tumour sample available (archival or recent biopsy), and no previous treatment with immunotherapy.

All participants will receive the study interventions of pembrolizumab and denosumab. All participants will receive the study interventions of pembrolizumab and denosumab. Pembrolizumab will be given every 3 weeks at a dose of 200mg and denosumab will be given on day 1, day 8, day 22 and then every 21 days (3 weekly) thereafter as a single subcutaneous injection. Treatment with pembrolizumab and denosumab will continue until evidence of clinical progression or prohibitive toxicity, or withdrawal of consent, up to a maximum duration of 2 years.

70 eligible participants will be recruited from 15 sites in Australia and New Zealand over a 2 year period.

ELIGIBILITY:
Inclusion Criteria:

* Adults, aged 18 years and older, with histologically confirmed unresectable or metastatic renal cell carcinoma with a clear cell component
* Disease progression during or after VEGFR TKI treatment
* At least 1 target lesion according to RECIST v1.1
* ECOG performance status of 0-2
* Adequate bone marrow function (done within 14 days prior to registration
* Haemoglobin ≥ 90g/L
* Platelet ≥ 75x109/L
* Neutrophil count ≥ 1.5x109/L
* Adequate liver function (done within 14 days prior to registration and with values within the ranges specified below):
* Bilirubin ≤ 1.5 x upper limit of normal (ULN) except for patients with known Gilbert's syndrome
* AST or ALT ≤ 3.0 x ULN (or ≤ 5.0x ULN in the presence of liver metastases)
* Adequate renal function (done within 14 days prior to registration and with values within the ranges specified below):
* Creatinine ≤ 1.5x ULN OR
* Creatinine clearance (CrCl) ≥ 30mL/min
* Serum calcium or albumin-adjusted serum calcium ≥2.0 mmol/L
* Tumour tissue available for tertiary correlative studies
* Willing and able to start treatment within 14 days of registration, and to comply with all study requirements, including the timing and/or nature of the required treatment and assessments
* Signed, written informed consent

Exclusion Criteria:

* Prior treatment with pembrolizumab, or with any other anti-PD-1, anti-PD-L1, Anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T cell co-stimulation or immune checkpoint pathways
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Any condition requiring systemic treatment with either corticosteroids (>10mg daily prednisone or equivalent dose of alternative corticosteroid) or other immunosuppressive medications within 14 days of pembrolizumab administration. Intranasal, inhaled or topical steroids are permitted in the absence of active autoimmune disease.
* Prior treatment with denosumab.
* Untreated brain or leptomeningeal metastases or current clinical or radiological progression of known brain metastases, or requirement for steroid therapy for brain metastases. Patients with treated brain metastases are eligible if they have been stable and off steroids for ≥ 3 weeks.
* Prior allogeneic organ transplant, inflammatory bowel disease, pneumonitis, tuberculosis, or primary immunodeficiency
* Active infection requiring systemic therapy within 14 days before the first dose of pembrolizumab
* Receipt of live attenuated vaccination within 30 days of the planned first dose of pembrolizumab
* Active dental or jaw condition that precludes administration of denosumab:

  i) Significant dental/oral disease, including prior history or current evidence of osteonecrosis/osteomyelitis of the jaw, or; ii) Active dental or jaw condition which requires oral surgery, or; iii) Non-healed dental/oral surgery, or; iv) Planned invasive dental procedures during the course of the study
* Clinically significant hypersensitivity to denosumab or any components of denosumab
* Targeted small molecule therapy, surgery or radiation therapy within 2 weeks before registration, or persisting adverse event(s) of Grade 2 or more due to a previously administered agent. Note that participants who have had recent major surgery must have recovered adequately before registration.
* Life expectancy of less than 3 months.
* History of an active malignancy within the previous 5 years, except for locally curable cancers that have been apparently cured, such as low-grade thyroid carcinoma, prostate cancer not requiring treatment (Gleason grade ≤ 6), basal or squamous cell skin cancer, superficial bladder cancer, melanoma in situ, or carcinoma in situ of the prostate, cervix, or breast. Patients who have been free of other malignancies for ≥ 5 years prior to registration are eligible for this study.
* Significant infection, including chronic active hepatitis B, hepatitis C, or HIV. - Serious medical or psychiatric conditions that might limit the ability of the patient to comply with the protocol
* Pregnancy, lactation, or inadequate contraception. Women must be post-menopausal, infertile, or use a reliable means of contraception. Women of childbearing potential must have a negative pregnancy test done within 7 days prior to registration. Men must have been surgically sterilised or use a (double if required) barrier method of contraception. Subject is excluded if pregnant or breast feeding, or planning to become pregnant within 5 months after the end of treatment. Female subject of child bearing potential is excluded if they are not willing to use, in combination with her partner, highly effective contraception during treatment and for 5 months after the end of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2023-06-04 (Estimated); Study Completion 2023-06-04 (Estimated)

PRIMARY OUTCOMES:
Objective tumour response | Through study completion, on average 3.5 years
  The objective tumour response rate, as assessed by RECIST1.1 - This is defined as the proportion of participants in the analysis set with a confirmed complete response (CR) or partial response (PR) divided by the number of participants in the analysis set.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 6 months
  Progression-free survival is defined as proportion alive and progression-free at 6 months, RECIST 1.1, iRECIST
Disease control rate (DCR) | 6 months
  Disease control rate is defined the proportion in CR, PR, or SD at 6 months iRECIST) rate (DCRR)
Time to objective tumour response (OTR) | Through study completion, on average 3.5 years
  Objective tumour response is defined as duration of OTR using RECIST 1.1 and iRECIST
Time to first skeletal related event (SRE) | Through study completion, on average 3.5 years
  This is defined as the interval from date of registration to the date of first evidence of first skeletal related event.
Frequency and severity of adverse events | From time of patient registration, until 100 days after the last dose of treatment
  The number of patients with adverse events, particularly immune-related adverse events, that are related to study drug, as assessed and graded according to CTCAE v4.03
Frequency of treatment delays and discontinuation due to toxicity | From time of patient registration, until 30 days after the last dose of treatment
  The number of participants with permanent discontinuation of treatment or delays due to toxicity, as assessed and graded according to CTCAE v4.03

OTHER OUTCOMES:
Identification of tumour markers to predict outcomes | Through study completion, on average 3.5 years
  Identifying tissue and circulating biomarkers that are prognostic and predictive of response to treatment, safety and resistance to study treatment (associations of biomarkers with clinical outcomes).

CONTACTS AND LOCATIONS:
Locations (16):
- Australia (16):
  - Border Medical Oncology Research Unit, Albury, New South Wales
  - Northern Cancer Institute, Frenchs Forest, New South Wales
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - St Vincent's Hospital Sydney, Sydney, New South Wales
  - St George, Sydney, New South Wales
  - Concord Repatriation General Hospital, Sydney, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Icon Cancer Care, Brisbane, Queensland
  - Royal Brisbane and Womens hospital, Herston, Queensland
  - Townsville Hospital, Townsville, Queensland
  - Flinders Medical Centre, Adelaide, South Australia
  - Box Hill, Box Hill, Victoria
  - Monash Health, Melbourne, Victoria
  - Peter MacCallum Cancer Center, Melbourne, Victoria
  - Ballarat Oncology & Haematology Services, Wendouree, Victoria
  - Fiona Stanley Hospital, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Within 12 months of study completion
Access Criteria: Authorised personnel as defined in the study contracts